CLINICAL TRIAL: NCT01273311
Title: Contribution of Diabetes and Its Causes to Signs of Brain Aging in a Young-to-Middle Age Cohort
Brief Title: CARDIA Brain MRI Substudy
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911071; 11-AG-N071
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-02-18

CONDITIONS: Brain Aging; Obesity; Diabetes
Keywords: Brain Aging; Diabetes; Aging; Obesity; CARDIA
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The Coronary Artery Risk Development in Young Adults (CARDIA) study is an investigation of cardiovascular risk factors among African-American and white young adults between 18 and 30 years of age, first recruited in 1985 86 from Birmingham, AL; Chicago, IL; Minneapolis, MN; and Oakland, CA. The study has examined a wide variety of risk factors, including insulin resistance, obesity, and diabetes. Based on 20 years of followup, the data provide evidence of an increase in the prevalence of many cardiovascular risk factors, as well as other factors that may lead to brain disease. To further evaluate these changes, the CARDIA Year 25 Exam will include a brain imaging component to study brain structure and function in a subset of CARDIA participants.

Objectives:

- To conduct brain magnetic resonance imaging as part of a 25-year followup study on participants in the original CARDIA study of heart disease risk factors in young adults.

Eligibility:

- Existing CARDIA study participants in the Minneapolis, MN, and Oakland, CA regions.

Design:

* Participants will be screened with a full medical history and physical examination. - Participants will have an MRI scan at the 25-year followup examination for the CARDIA study.
* No additional testing or treatment will be required for this protocol.

DETAILED DESCRIPTION:
The Coronary Artery Risk Development in Young Adults (CARDIA) Study is a prospective, epidemiologic investigation of the determinants and evolution of cardiovascular risk factors among 5,115 African American and white young to middle age adults 18-30 years of age at baseline in 1985-86. Participants were recruited from the populations of four geographic locations (Birmingham, AL; Chicago, IL; Minneapolis, MN; and Oakland, CA). The study population was approximately balanced according to sex (54% women), ethnicity (52% African American), and education (40% with less than equal to 12 years of education) at each center (Friedman). After the 1984 baseline, additional examinations were undertaken at years 2 (1987-88), 5 (1990-91), 7 (1992-93), 10 (1995-96), 15 (2000-01) and 20 (2005-06). To date, 72% of the total baseline cohort is still active in the study.

Based on 20 years of follow-up, the longitudinal data on this cohort provide clear evidence of an increase in the prevalence of many cardiovascular risk factors, including obesity and diabetes. Therefore, the study presents an ideal and unique opportunity to study change in cardiovascular risk factors beginning at an age we hypothesize may be critical in determining future trajectories of brain disease. Furthermore, the trends in CV-RF reflect general trends in the US population. Thus, CARDIA participants are ideal to study now because the cohort reflects the characteristics of the next generation of older persons.

This is an ancillary study of MRI-evident neurodegenerative and vascular brain changes in a subset of 719 CARDIA participants who participate in the Year 25 Exam. Specifically, we will study the relations of timing length of exposure and levels of cardiovascular risk factors to presence of sub-clinical brain lesions and cognitive impairments. Participants were recruited from the CARDIA field sites at Birmingham, AL (PI: Cora E. Lewis, MD, MSPH- University of Lalbama, Nirmingham), Minneapolis, MN (PI: Pamela Schreiner, PhD, MS- University of Minnesota) and Oakland, CA (PI: Steve Sidney, MD, mPH- Kaiser Permanente).

ELIGIBILITY:
* INCLUSION CRITERIA:

A qualified participant from the CARDIA trial that does not have any of the below MRI contraindications.

EXCLUSION CRITERIA:

Participants with a known contraindication to an MRI examination will be excluded from the study (severe claustrophobia, pacemaker, defibrillator, neuro-stimulator, ferro-magnetic aneurysm clip or an unknown, 3T MR incompatible metal implant of any kind or any foreign metal objects in the body such as bullets, shrapnel, metal slivers, etc).

Any female participant of childbearing age who has not tested negative on a pregnancy test prior to the scheduled MRI exam will also be excluded from participation in the Brain MRI Substudy.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 719 (Actual)
Dates: Start 2010-12-22; Study Completion 2014-02-18

CONTACTS AND LOCATIONS:
Overall Officials: Lenore J Launer, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Friedman GD, Cutter GR, Donahue RP, Hughes GH, Hulley SB, Jacobs DR Jr, Liu K, Savage PJ. CARDIA: study design, recruitment, and some characteristics of the examined subjects. J Clin Epidemiol. 1988;41(11):1105-16. doi: 10.1016/0895-4356(88)90080-7. PMID 3204420
- [Background] Mainous AG 3rd, Baker R, Koopman RJ, Saxena S, Diaz VA, Everett CJ, Majeed A. Impact of the population at risk of diabetes on projections of diabetes burden in the United States: an epidemic on the way. Diabetologia. 2007 May;50(5):934-40. doi: 10.1007/s00125-006-0528-5. Epub 2006 Nov 21. PMID 17119914